CLINICAL TRIAL: NCT05370183
Title: Tenotomy of Biceps' Long Head by Mini-optics in Consultation (Hyperambulatory): What Advantage Compared to the Operating Room?
Acronym: NANOBICEPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-AOI-13
Record Dates: First submitted 2022-04-29; First posted 2022-05-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Pain; Biceps Tendon Disorder
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperambulatory tenotomy (Experimental): regarding randomization result, patient wil have a tenotomy of biceps' long head by mini-optics in consultation
  Interventions: Procedure: Hyperambulatory tenotomy
- Operating room tenotomy (Active Comparator): regarding randomization result, patient wil have a tenotomy of biceps' long head upon arthroscopy under normal operating condition
  Interventions: Procedure: Operating room tenotomy

INTERVENTIONS:
Procedure: Hyperambulatory tenotomy — Using mini-optics a minimally invasive device, hypermabulatory tenotomy is performed in consultation, with a local anethesia
  Arms: Hyperambulatory tenotomy
Procedure: Operating room tenotomy — Operating room tenotomy is performed according standard practice, with general anesthesia.
  Arms: Operating room tenotomy

SUMMARY:
Mini-optics has been used in orthopedics for a short time. The Nanoscope used in this study is marketed by Arthrex. Its main indications concern knee, elbow, wrist, carp and small joints of long fingers for diagnostic and sometimes therapeutic purposes. Some teams use it to replace expensive radiological examinations and/or difficult to access, in consultation, for diagnostic in the knee, but also for therapeutic for partial meniscectomy with several related publications. The investigators recently published a feasibility study of isolated tenotomy of the biceps with this minimally invasive device in consultation (first indexed article describing this technique).

This project is part of the broader context of "In Office" surgery, for which there are many applications. Through the miniaturisation of optics and access to "portable" technologies, surgical procedures can now be performed in consultation ("In Office"). For example: release of the carpal tunnel or ulnar canal to the elbow under ultrasound, partial meniscectomy, removal of foreign body from the elbow in consultation.

Indeed, in addition to the technical interest of this innovation for a simple and frequent surgical procedure, it should make it possible to transpose anxiety management for the patient, time-consuming and costly for the institution into a heavy technical platform (operating room) towards a simplified, fast and streamlined approach in consultation. In the scientific literature, other equivalent surgical procedures have already been identified and performed in consultation with various tools (carpal tunnel, ulnar nerve in the elbow, meniscectomy in the knee but also in other surgical specialties such as cataract in ophthalmology) with better patient satisfaction, improved patient journey, reduced costs, an increase in the number of patients treated.

The investigators wish to demonstrate the non-inferiority of intraarticular tenotomy of the biceps long head performed in consultation with mini-optics and local anaesthesia compared to the operating room in order to modify practices and optimize the management of patients within the institution while improving their satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 years-old,
* With shoulder pain associated to massive irreparable rotator cuff and a biceps still presents (premature Hamada's stages, 1 to 3); Or with an isolated pathology of biceps with intact rotator cuff (in particular bicipital instability, subluxation, tenosynovitis, pre-rupture)
* Indication for tenotomy according orthopedic surgeon
* having given written consent after written and oral information,
* member of the social security system.

Exclusion Criteria:

* patient protected by law or under guardianship r curatorship, or not able to participae in a clinical trial under L.1121-16 article of French Public Health Regulations
* pregnant or nursing patient,
* Allergies to local anesthetics
* Athletes
* Capsulitis in progress
* history of shoulder surgery
* Medical history of infection
* fracture of proximal end of the humerus
* Patient refusal to take part

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on pain felt by patient | At inclusion (V0)
  Pain felt will be assessed with a visual and analog scale for pain. The scale ranges from 0 (no pain) to 10 (maximum thinkable pain). Limit of non-inferiority is fixed to 1.5 on this scale.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on pain felt by patient | 3 hours after surgery (V1)
  Pain felt will be assessed with a visual and analog scale for pain. The scale ranges from 0 (no pain) to 10 (maximum thinkable pain). Limit of non-inferiority is fixed to 1.5 on this scale.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on pain felt by patient | The day after surgery (V2)
  Pain felt will be assessed with a visual and analog scale for pain. The scale ranges from 0 (no pain) to 10 (maximum thinkable pain). Limit of non-inferiority is fixed to 1.5 on this scale.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on pain felt by patient | 2 weeks after surgery (V3)
  Pain felt will be assessed with a visual and analog scale for pain. The scale ranges from 0 (no pain) to 10 (maximum thinkable pain). Limit of non-inferiority is fixed to 1.5 on this scale.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on pain felt by patient | 6 weeks after surgery (V4)
  Pain felt will be assessed with a visual and analog scale for pain. The scale ranges from 0 (no pain) to 10 (maximum thinkable pain). Limit of non-inferiority is fixed to 1.5 on this scale.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on pain felt by patient | 3 months after surgery (V5)
  Pain felt will be assessed with a visual and analog scale for pain. The scale ranges from 0 (no pain) to 10 (maximum thinkable pain). Limit of non-inferiority is fixed to 1.5 on this scale.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on pain felt by patient | 6 months after surgery (V6)
  Pain felt will be assessed with a visual and analog scale for pain. The scale ranges from 0 (no pain) to 10 (maximum thinkable pain). Limit of non-inferiority is fixed to 1.5 on this scale.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on pain felt by patient | 12 months after surgery (V7)
  Pain felt will be assessed with a visual and analog scale for pain. The scale ranges from 0 (no pain) to 10 (maximum thinkable pain). Limit of non-inferiority is fixed to 1.5 on this scale.

SECONDARY OUTCOMES:
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on number of scare | 2 weeks (V3) after surgery
  Number of scare will be visually evaluated by investigators
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on number of scare | 6 weeks (V4) after surgery
  Number of scare will be visually evaluated by investigators
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on number of scare | 3 months (V5) after surgery
  Number of scare will be visually evaluated by investigators
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on number of scare | 6 months (V6) after surgery
  Number of scare will be visually evaluated by investigators
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on number of scare | 12 months (V7) after surgery
  Number of scare will be visually evaluated by investigators
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on scare's length | 2 weeks (V3) after surgery
  Scare's length will be assessed by investigator with a small ruler, in millimeter.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on scare's length | 6 weeks after surgery
  Scare's length will be assessed by investigator with a small ruler, in millimeter.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on scare's length | 3 months (V5) after surgery
  Scare's length will be assessed by investigator with a small ruler, in millimeter.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on scare's length | 6 months (V6) after surgery
  Scare's length will be assessed by investigator with a small ruler, in millimeter.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on scare's length | 12 months (V7) after surgery
  Scare's length will be assessed by investigator with a small ruler, in millimeter.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on scare's width | 2 weeks (V3) after surgery
  Scare's width will be assessed by investigator with a small ruler, in millimeter.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on scare's width | 6 weeks (V4) after surgery
  Scare's width will be assessed by investigator with a small ruler, in millimeter.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on scare's width | 3 months (V5) after surgery
  Scare's width will be assessed by investigator with a small ruler, in millimeter.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on scare's width | 6 months (V6) after surgery
  Scare's width will be assessed by investigator with a small ruler, in millimeter.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on scare's width | 12 months (V7) after surgery
  Scare's width will be assessed by investigator with a small ruler, in millimeter.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on time to onset | 2 weeks (V3) after surgery
  Time to onset will be evaluated by investigator, in number of days.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on time to onset | 6 weeks (V4) after surgery
  Time to onset will be evaluated by investigator, in number of days.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on time to onset | 3 months (V5) after surgery
  Time to onset will be evaluated by investigator, in number of days.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on time to onset | 6 months (V6) after surgery
  Time to onset will be evaluated by investigator, in number of days.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality, in particular on time to onset | 12 months (V7) after surgery
  Time to onset will be evaluated by investigator, in number of days.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality,in particular on possible desunion | 2 weeks (V3) after surgery
  Desunion will be evaluated by investigator, with 2 possible values : yes or no.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality,in particular on possible desunion | 6 weeks (V4) after surgery
  Desunion will be evaluated by investigator, with 2 possible values : yes or no.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality,in particular on possible desunion | 3 months (V5) after surgery
  Desunion will be evaluated by investigator, with 2 possible values : yes or no.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality,in particular on possible desunion | 6 months (V6) after surgery
  Desunion will be evaluated by investigator, with 2 possible values : yes or no.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on scare quality,in particular on possible desunion | 12 months (V7) after surgery
  Desunion will be evaluated by investigator, with 2 possible values : yes or no.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on shoulder function, in particular on active and passive mobility | At inclusion (V0)
  Active and passive mobility of both shoulders will be assessed by investigator on following parameters: abduction, adduction, flexion extension, internal and external rotation. All theses paramèters will be assessed with a goniometer, in degree.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on shoulder function, in particular on active and passive mobility | 2 weeks (V3) after surgery
  Active and passive mobility of both shoulders will be assessed by investigator on following parameters: abduction, adduction, flexion extension, internal and external rotation. All theses paramèters will be assessed with a goniometer, in degree.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on shoulder function, in particular on active and passive mobility | 6 weeks (V4) after surgery
  Active and passive mobility of both shoulders will be assessed by investigator on following parameters: abduction, adduction, flexion extension, internal and external rotation. All theses paramèters will be assessed with a goniometer, in degree.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on shoulder function, in particular on active and passive mobility | 3 months (V5) after surgery
  Active and passive mobility of both shoulders will be assessed by investigator on following parameters: abduction, adduction, flexion extension, internal and external rotation. All theses paramèters will be assessed with a goniometer, in degree.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on shoulder function, in particular on active and passive mobility | 6 months (V6) after surgery
  Active and passive mobility of both shoulders will be assessed by investigator on following parameters: abduction, adduction, flexion extension, internal and external rotation. All theses paramèters will be assessed with a goniometer, in degree.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on shoulder function, in particular on active and passive mobility | 12 months (V7) after surgery
  Active and passive mobility of both shoulders will be assessed by investigator on following parameters: abduction, adduction, flexion extension, internal and external rotation. All theses paramèters will be assessed with a goniometer, in degree.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on shoulder function, in particular on Subjective Shoulder Value | At inclusion (V0)
  The Subjective Shoulder Value will be evalued by patient himself, by answering the following question: What value do you give to your shoulder, out of 100, compared to a normal shoulder rated at 100% ? this scale ranges from 0 (non-functional shoulder) to 100 (normal shoulder)
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on shoulder function, in particular on Subjective Shoulder Value | 2 weeks (V3) after surgery
  The Subjective Shoulder Value will be evalued by patient himself, by answering the following question: What value do you give to your shoulder, out of 100, compared to a normal shoulder rated at 100% ? this scale ranges from 0 (non-functional shoulder) to 100 (normal shoulder)
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on shoulder function, in particular on Subjective Shoulder Value | 6 weeks (V4) after surgery
  The Subjective Shoulder Value will be evalued by patient himself, by answering the following question: What value do you give to your shoulder, out of 100, compared to a normal shoulder rated at 100% ? this scale ranges from 0 (non-functional shoulder) to 100 (normal shoulder)
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on shoulder function, in particular on Subjective Shoulder Value | 3 months (V5) after surgery
  The Subjective Shoulder Value will be evalued by patient himself, by answering the following question: What value do you give to your shoulder, out of 100, compared to a normal shoulder rated at 100% ? this scale ranges from 0 (non-functional shoulder) to 100 (normal shoulder)
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on shoulder function, in particular on Subjective Shoulder Value | 6 months (V6) after surgery
  The Subjective Shoulder Value will be evalued by patient himself, by answering the following question: What value do you give to your shoulder, out of 100, compared to a normal shoulder rated at 100% ? this scale ranges from 0 (non-functional shoulder) to 100 (normal shoulder)
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on shoulder function, in particular on Subjective Shoulder Value | 12 months (V7) after surgery
  The Subjective Shoulder Value will be evalued by patient himself, by answering the following question: What value do you give to your shoulder, out of 100, compared to a normal shoulder rated at 100% ? this scale ranges from 0 (non-functional shoulder) to 100 (normal shoulder)
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on patient satisfaction, with Constant's score | At inclusion (V0)
  Patient satisfaction will be evaluated using Constant's score, a quantitative value from 0 to 100.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on patient satisfaction, with Constant's score | 2 weeks (V3) after surgery
  Patient satisfaction will be evaluated using Constant's score, a quantitative value from 0 to 100.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on patient satisfaction, with Constant's score | 6 weeks (V4) after surgery
  Patient satisfaction will be evaluated using Constant's score, a quantitative value from 0 to 100.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on patient satisfaction, with Constant's score | 3 months (V5) after surgery
  Patient satisfaction will be evaluated using Constant's score, a quantitative value from 0 to 100.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on patient satisfaction, with Constant's score | 6 months (V6) after surgery
  Patient satisfaction will be evaluated using Constant's score, a quantitative value from 0 to 100.
Demonstrate the non-inferiority of tenotomy of biceps' long head by mini-optics in consultation (hyperambulatory) compared to upon arthroscopy under normal operating condition on patient satisfaction, with Constant's score | 12 months (V7) after surgery
  Patient satisfaction will be evaluated using Constant's score, a quantitative value from 0 to 100.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, Alpes Maritimes, France

IPD SHARING:
Plan to Share IPD: No